CLINICAL TRIAL: NCT04535388
Title: Efficacy and Safety of LK Scleral Lens for Patients With Intractable Ocular Surface Diseases: A Prospective, Multicenter, Open-Label, Single-Arm Clinical Trial
Brief Title: LK Scleral Lens for Patients With Intractable Ocular Surface Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LK Scleral Lens
Record Dates: First submitted 2020-08-18; First posted 2020-09-02 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-08

CONDITIONS: Ocular Surface Disease
Keywords: Cornea; LK scleral lens; Ocular surface disease; Scleral lens
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LK scleral lens (Other): LK scleral lens (Lucid Korea LTD, Seoul, Republic of Korea) are worn for 12 weeks.
  Interventions: Device: LK scleral lens

INTERVENTIONS:
Device: LK scleral lens — LK scleral lens fitting and application were done for 12 weeks.

SUMMARY:
Scleral lenses have emerged as an efficacious treatment option for various types of intractable ocular surface diseases with many advantageous results. The purpose of this study was to report the efficacy and safety of the LK scleral lenses and determine their suitability in Asian patients with intractable ocular surface diseases. Subjects with intractable ocular surface diseases are enrolled to fit LK scleral lenses for 12 weeks for a prospective study. Evaluations are performed at 1, 4, 8 and 12 weeks. General patient demographics and medical history, visual acuities, thorough ophthalmic evaluation, ocular surface disease index and National Eye Institute 25-Item Visual Function Questionnaire are collected for each patient.

DETAILED DESCRIPTION:
To date, there are several commercially manufactured scleral lenses of different designs and sizes, all of which have been proven to be clinically beneficial in a wide spectrum of diseases. Especially in the management of intractable ocular surface diseases, scleral lenses with large diameters are commonly used so that the lens entirely rests on the sclera with sufficient tear reservoir. PROSE devices (Boston Foundation for Sight, Needham, MA), one of the first and representative scleral lenses shown to have long-term clinical benefits for complex corneal diseases, have large diameters of 17.5 to 23.0 mm. However, in Republic of Korea, only scleral lenses with small diameters are currently available. SoClearⓇ and OnefitⓇ scleral lenses, two of the most commonly used scleral lenses in Republic of Korea, possess diameters ranging from 14.1 to 15.5 mm and 13.3 to 15.0 mm, respectively, and are not actually fully scleral but more of a corneoscleral type lenses. Furthermore, Asians have smaller palpebral fissures with tighter eyelids than the Western population, which may restrict patients' tolerability of wearing a large scleral lens and limit its clinical benefits. Therefore, a more suitable scleral lens for Asians with larger diameter is required.

Accordingly, this study investigates the efficacy and safety of the LK scleral lens (Lucid Korea LTD, Seoul, Republic of Korea), which has been newly manufactured to have larger diameters than currently available commercial lenses, and determines their suitability in Asian patients with intractable ocular surface diseases.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 to 69 years
* Intractable ocular surface disease
* Uncorrected visual acuity better than count finger and ≥ 0.3 logMAR (log of the Minimum Angle of Resolution)
* Best-corrected visual acuity ≥ 0.3 logMAR (log of the Minimum Angle of Resolution)

Exclusion Criteria:

* Currently under treatment for infectious keratitis
* Difficulty of scleral lens application due to severe allergic conjunctivitis, low compliance, and other potential contraindications
* Diabetes mellitus and/or hypertension
* Pregnant or planning pregnancy E. Unwilling to follow study schedule F. Enrolled in another clinical study G. Determined inappropriate under investigators' discretion

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2014-03-31 (Actual); Study Completion 2014-04-22 (Actual)

PRIMARY OUTCOMES:
Change of visual improvement after wearing the LK scleral lens | Change from baseline best corrected visual acuity at week 1
  Best corrected visual acuity is measured. Snellen visual acuity is converted to log of the Minimum Angle of Resolution for assessment.
Change of visual improvement after wearing the LK scleral lens | Change from baseline best corrected visual acuity at week 4
  Best corrected visual acuity is measured. Snellen visual acuity is converted to log of the Minimum Angle of Resolution for assessment.
Change of visual improvement after wearing the LK scleral lens | Change from baseline best corrected visual acuity at week 8
  Best corrected visual acuity is measured. Snellen visual acuity is converted to log of the Minimum Angle of Resolution for assessment.
Change of visual improvement after wearing the LK scleral lens | Change from baseline best corrected visual acuity at week 12
  Best corrected visual acuity is measured. Snellen visual acuity is converted to log of the Minimum Angle of Resolution for assessment.
Change of ocular surface state after wearing the LK scleral lens | Change from baseline ocular surface state at week 1
  0.5% Fluorescein application to the ocular surface and observation under blue light exhibits ocular surface epithelial erosions that are associated with chronic dry eyes and irregular tear film status. Grading is performed through Oxford Grading which ranges from 0 = none to 5 = severe.
Change of ocular surface state after wearing the LK scleral lens | Change from baseline ocular surface state at week 4
  0.5% Fluorescein application to the ocular surface and observation under blue light exhibits ocular surface epithelial erosions that are associated with chronic dry eyes and irregular tear film status. Grading is performed through Oxford Grading which ranges from 0 = none to 5 = severe.
Change of ocular surface state after wearing the LK scleral lens | Change from baseline ocular surface state at week 8
  0.5% Fluorescein application to the ocular surface and observation under blue light exhibits ocular surface epithelial erosions that are associated with chronic dry eyes and irregular tear film status. Grading is performed through Oxford Grading which ranges from 0 = none to 5 = severe.
Change of ocular surface state after wearing the LK scleral lens | Change from baseline ocular surface state at week 12
  0.5% Fluorescein application to the ocular surface and observation under blue light exhibits ocular surface epithelial erosions that are associated with chronic dry eyes and irregular tear film status. Grading is performed through Oxford Grading which ranges from 0 = none to 5 = severe.
Change of subjective ocular surface discomfort after wearing the LK scleral lens | Change from baseline 25-Item Visual Function Questionnaire scores at week 1
  25-Item Visual Function Questionnaire scores is a validated self-reporting dry eye symptom questionnaires. The scores are graded from 0 = no symptoms to 100 = all symptoms with the most severity.
Change of subjective ocular surface discomfort after wearing the LK scleral lens | Change from baseline 25-Item Visual Function Questionnaire scores at week 4
  25-Item Visual Function Questionnaire scores is a validated self-reporting dry eye symptom questionnaires. The scores are graded from 0 = no symptoms to 100 = all symptoms with the most severity.
Change of subjective ocular surface discomfort after wearing the LK scleral lens | Change from baseline 25-Item Visual Function Questionnaire scores at week 8
  25-Item Visual Function Questionnaire scores is a validated self-reporting dry eye symptom questionnaires. The scores are graded from 0 = no symptoms to 100 = all symptoms with the most severity.
Change of subjective ocular surface discomfort after wearing the LK scleral lens | Change from baseline 25-Item Visual Function Questionnaire scores at week 12
  25-Item Visual Function Questionnaire scores is a validated self-reporting dry eye symptom questionnaires. The scores are graded from 0 = no symptoms to 100 = all symptoms with the most severity.
Change of subjective ocular surface discomfort after wearing the LK scleral lens | Change from baseline ocular surface disease index at week 1
  Ocular surface disease index is validated self-reporting dry eye symptom questionnaires. The scores are graded from 0 = no symptoms to 48 = all symptoms with the most severity.
Change of subjective ocular surface discomfort after wearing the LK scleral lens | Change from baseline ocular surface disease index at week 4
  Ocular surface disease index is validated self-reporting dry eye symptom questionnaires. The scores are graded from 0 = no symptoms to 48 = all symptoms with the most severity.
Change of subjective ocular surface discomfort after wearing the LK scleral lens | Change from baseline ocular surface disease index at week 8
  Ocular surface disease index is validated self-reporting dry eye symptom questionnaires. The scores are graded from 0 = no symptoms to 48 = all symptoms with the most severity.
Change of subjective ocular surface discomfort after wearing the LK scleral lens | Change from baseline ocular surface disease index at week 12
  Ocular surface disease index is validated self-reporting dry eye symptom questionnaires. The scores are graded from 0 = no symptoms to 48 = all symptoms with the most severity.
Adverse effects after wearing the LK scleral lens | Week 12
  Scleral lenses can cause endothelial cell density decrease and corneal edema. Endothelial cell density was assessed using a noncontact specular microscope, while corneal edema whereabouts was evaluating corneal thickness using ultrasound pachymetry.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moon J, Lee SM, Hyon JY, Kim MK, Oh JY, Choi HJ. Large diameter scleral lens benefits for Asians with intractable ocular surface diseases: a prospective, single-arm clinical trial. Sci Rep. 2021 Jan 27;11(1):2288. doi: 10.1038/s41598-021-82010-z. PMID 33504920